CLINICAL TRIAL: NCT00978432
Title: A Phase 2 Study to Evaluate the Efficacy of Epigenetic Modulation in Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Epigenetic Modulation in Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The toxicity seemed to outweigh the benefit.
Sponsor: Anne Beaven, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Anne Beaven, MD, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012947
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: NHL; DLBCL; recurrent; refractory; de novo
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Everolimus; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1a (RAD001 followed by LBH589) (Experimental): Part 1a: Sequential single agent therapy with RAD001 and LBH589. Each agent will be given for four-six 28-day cycles.
  Subjects with less than a CR after 4 cycles of study drug should proceed to the next study drug(s) after the prescribed washout period.
  Subjects with a CR may receive up to 6 cycles of study drug and will not receive the next study drug(s) until there is evidence of progressive disease.
  There will be a 1-6 week 'washout' period between stopping and starting each agent in Part 1, unless rapid progression suggests holding therapy would not be in the patient's best interest.
  Interventions: Drug: RAD001; Drug: LBH589
- Arm 1b (LBH589 followed by RAD001) (Experimental): Part 1b: Sequential single agent therapy with LBH589 and RAD001 . Each agent will be given for four-six 28-day cycles.
  Subjects with less than a CR after 4 cycles of study drug should proceed to the next study drug(s) after the prescribed washout period.
  Subjects with a CR may receive up to 6 cycles of study drug and will not receive the next study drug(s) until there is evidence of progressive disease.
  There will be a 1-6 week 'washout' period between stopping and starting each agent in Part 1, unless rapid progression suggests holding therapy would not be in the patient's best interest.
  Interventions: Drug: RAD001; Drug: LBH589
- Doublet (Combination RAD001 and LBH589) (Experimental): Subjects will receive the doublet of RAD001 and LBH589 given in two to thirteen, 28-day cycles. Subjects will be evaluated for the disease status after completion of cycle two and then after every 4 cycles. Subjects with progressive disease will stop after 2 cycles. Subjects with stable disease or better may receive up to 13 cycles. LBH589 will start at 15mg po three days a week at least 2 days apart such as on days M/W/F or T/Th/Sat and RAD001 will start at 7.5mg po daily.
  Interventions: Drug: Doublet (RAD001 and LBH589)

INTERVENTIONS:
Drug: RAD001 — 10 mg/day for Part 1 of the trial
  Other Names: Everolimus
  Arms: Arm 1a (RAD001 followed by LBH589); Arm 1b (LBH589 followed by RAD001)
Drug: LBH589 — 40 mg on Monday, Wednesday and Friday weekly for Part 1 of the trial
  Other Names: panobinostat
  Arms: Arm 1a (RAD001 followed by LBH589); Arm 1b (LBH589 followed by RAD001)
Drug: Doublet (RAD001 and LBH589) — RAD001 7.5 mg by mouth daily and LBH589 15 mg by mouth on Monday/Wednesday/Friday during Part 2.
  Arms: Doublet (Combination RAD001 and LBH589)

SUMMARY:
The purpose of this study is evaluate the response, safety and tolerability in subjects receiving the investigational drugs, RAD001 and LBH589. Subjects in Part 1 will receive one drug for four cycles followed by 4 cycles of the second drug unless they achieve complete remission. Subjects in a complete remission may receive up to 6 cycles of study drug and will not receive the next study drug until there is evidence of disease progression. Subjects in Part 2 will receive both drugs together for at least 2 cycles and up to 13 if tolerated.

DETAILED DESCRIPTION:
This will be a prospective, non-randomized, un-blinded phase 2 efficacy trial using a mechanistic target of rapamycin (mTOR) inhibitor and a histone deacetylase (HDAC) inhibitor for epigenetic targeted therapies.

Subjects will receive RAD001 and LBH589 given in two to thirteen, 28-day cycles. Subjects will be assessed for disease status after 2 cycles and then after every 4 cycles. Subjects with progressive disease will stop after 2 cycles. Subjects with stable disease or better les may receive up to 13 cycles. LBH589 was given at 40mg when the study first opened and was changed to 20mg po shortly thereafter. LBH589 is taken on days M/W/F. RAD001 was given at 10mg po daily for Part 1. In Part 2, LBH589 is given at 15mg and RAD001 is given at 7.5mg.

Treatment will be administered on an outpatient basis. Patients will be followed for up to 2 years after completion of therapy or until progression of disease or death.

ELIGIBILITY:
Inclusion Criteria:

1. de novo or transformed Diffuse large B cell non-Hodgkin lymphoma (DLBCL). DLBCL-like lymphomas allowed:

   * Epstei-Barr virus (EBV)+ DLBCL in elderly,
   * DLBCL with chronic inflammation,
   * Primary cutaneous DLBCL, leg type,
   * B cell lymphoma unclassifiable - between DLBCL and Burkitt lymphoma,
   * B cell lymphoma unclassifiable - between large B cell lymphoma and classical Hodgkin lymphoma,
   * Anaplastic lymphoma kinase (ALK)+ large B cell lymphoma,
   * T cell histiocyte rich large B cell lymphoma
   * Primary mediastinal B cell lymphoma
   * Follicular grade 3 B cell lymphoma
2. Refractory or relapsed disease to >/= 1 prior treatment regimen: should include autologous stem cell transplant unless patient refused or ineligible.
3. Age > 18 years old
4. Eastern Cooperative Oncology Group (ECOG) performance status <2.
5. Measurable or evaluable disease by physical exam, radiographs or bone marrow involvement
6. Frozen tumor or paraffin-embedded sample available.
7. 3-4 core fresh/fresh-frozen biopsy specimens available. Leukapheresis may be done for patients with leukocytosis.
8. Laboratory Values per protocol.

Exclusion Criteria:

1. Laboratory Values

   * Grade 3 hyperlipidemia (Serum cholesterol >400mg/dl or serum triglycerides >5 x ULN)
   * Serum Glucose > 250mg/dl on >/= 2 checks on 2 separate days
   * Diabetics accepted if sugars controlled
2. Unlimited prior chemotherapy regimens, however:

   * No prior exposure to RAD001 or LBH589 or drugs that target mTOR (sirolimus, temsirolimus, etc) or HDAC (vorinostat)

     * No valproic acid during study or 5 days preceding start of first drug
   * No chemotherapy, biologics or immunotherapy < 2 weeks before registration (6 weeks if last received bis-chloroethylnitrosourea (BCNU) or mitomycin C). Subjects must be recovered from therapy-related non-hematological toxicities to < grade 1 or baseline if started with > grade 1 toxicity.
   * No time limit for radiation prior to registration.
   * No radioimmunotherapy < 2 months prior to registration. Subjects must be recovered from therapy-related toxicities to < grade 1 or baseline if started with > grade 1 toxicity.
   * No prior allogeneic stem cell transplantation unless allogeneic engraftment is <2%.
   * Subjects receiving chronic, systemic treatment with corticosteroids = to >20mg of prednisone per day.

     * Subjects receiving replacement for adrenal insufficiency allowed.
     * Topical or inhaled corticosteroids allowed.
3. History of other primary malignancy < 3 years ago, except inactive basal, squamous cell carcinoma of the skin or superficial melanoma only requiring excision, prostate cancer with a prostate specific antigen (PSA) stable for >/=3 months, carcinoma in situ of cervix.
4. Major surgery < 4 weeks before or Minor surgery < 2 weeks before registration. Subjects must be recovered from toxicities to < grade 1 or baseline if started with > grade 1 toxicity.
5. Investigational drugs < 4 weeks prior to registration.
6. Impaired Cardiac Function per protocol.
7. Pregnant or breastfeeding females or adults of reproductive potential not using effective birth control
8. Diffusing capacity or transfer factor of the lung for carbon monoxide (DLCO) < 40% if tested (per protocol).
9. Impaired lung function: O2 saturation 88% or less at rest on room air by Pulse Oximetry.
10. Immunization with live attenuated vaccines < 1 week of study entry
11. Impaired GI function or GI disease that may alter absorption of RAD001 or LBH589
12. Concurrent severe &/or uncontrolled medical conditions
13. Medications with risk of prolonging QT interval or inducing torsade de pointes or interacting with LBH589 and RAD001 may be used per the protocol.
14. Active bleeding tendency
15. Positive for HIV.
16. Positive for Hepatitis C virus (HCV).
17. History of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne W. Beaven, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment in October, 2009. 50 subjects were consented until enrollment closure in April 2015. Patients were recruited at the Duke Cancer Center Hematology clinic.
Pre-assignment Details: Fifty (50) participants signed consent. Eleven subjects were screen failures. The PI removed three subjects prior to treatment to receive alternate therapy. Three subjects chose to withdraw from the study prior to treatment.
Groups:
- Arm 1a (RAD001 Followed by LBH589): Part 1a: Sequential single agent therapy with RAD001 and LBH589. Each agent will be given for four-six 28-day cycles.
  Subjects with less than a CR after 4 cycles of study drug should proceed to the next study drug(s) after the prescribed washout period.
  Subjects with a CR may receive up to 6 cycles of study drug and will not receive the next study drug(s) until there is evidence of progressive disease.
  There will be a 1-6 week 'washout' period between stopping and starting each agent in Part 1, unless rapid progression suggests holding therapy would not be in the patient's best interest.
  RAD001: 10 mg/day for Part 1 of the trial
  LBH589: 40 mg on Monday, Wednesday and Friday weekly for Part 1 of the trial
- Arm 1b (LBH589 Followed by RAD001): Part 1b: Sequential single agent therapy with LBH589 and RAD001 . Each agent will be given for four-six 28-day cycles.
  Subjects with less than a CR after 4 cycles of study drug should proceed to the next study drug(s) after the prescribed washout period.
  Subjects with a CR may receive up to 6 cycles of study drug and will not receive the next study drug(s) until there is evidence of progressive disease.
  There will be a 1-6 week 'washout' period between stopping and starting each agent in Part 1, unless rapid progression suggests holding therapy would not be in the patient's best interest.
  RAD001: 10 mg/day for Part 1 of the trial
  LBH589: 40 mg on Monday, Wednesday and Friday weekly for Part 1 of the trial
Period: Overall Study
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Started | 10 | 5 | 18
Completed | 7 | 4 | 13
Not Completed | 3 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 3
Not completed — Adverse Event | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589) | Total
Number analyzed (Participants) | 10 | 5 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 9 | 16
  >=65 years | 5 | 3 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 3 | 10
  Male | 4 | 4 | 15 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 9 | 5 | 17 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate is the number of participants with a partial and complete response assessed by the Updated Cheson criteria for lymphoma. A complete response is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy and normalization of those biochemical abnormalities. If a subject has residual lesions on CT scan and the disease was fluorodeoxyglucose (FDG) avid pre-treatment, then that subject will be considered to be in a complete response. Partial response is a greater than or equal to 50% decrease in the sum of the products of the greatest diameters of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease
Time Frame: after 2 cycles of each study drug or after 2 cycles of doublet, up to 24 weeks
Population: Patients have to be on each drug for at least 2 cycles to be evaluable for response.
Measure: Number; unit: participants
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Number analyzed (Participants) | 10 | 5 | 18
participants | 1 | 0 | 4

2. Primary Outcome: Assessment of Association Between Observed Response to RAD001 and LBH589 and the Response Predicted by Molecular Signatures Developed in Our Pre-clinical Model
Description: We will estimate the association of the molecular signature-predicted response to the doublet (CR+PR) with the observed response. All evaluable patients will be used in estimating response. The chi-square test with one-sided alpha of 0.10 will be used to test for the association between predicted and observed responses. Contingency tables will be used to present these associations.
Time Frame: From the start of combination therapy until a maximum of 2 years after completion of therapy
Population: The number of responses to treatment were so few that we did not think we could get enough meaningful data for analysis. Therefore, molecular analysis was not performed and no results are available.
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Summary of Adverse Events (AEs)
Description: Counts of adverse events or treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose) experienced by patients on study drug(s). National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) is used to assess severity. Relatedness to study drug is assessed by the investigator.
Time Frame: From the time of first dose of study drug until 4 weeks after participant has stopped study drug; up to 1 year
Population: Participants who consented to the study and took study drug were analyzed for this outcome measure. Total number of events per CTCAE v4 category per arm are reported if more than one event occurred.
Measure: Number; unit: events
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Number analyzed (Participants) | 10 | 5 | 18
events
  Blood and lymphatic AEs | 18 | 6 | 42
  Gastrointestinal AEs | 30 | 10 | 39
  General Disorder AEs | 6 | 5 | 19
  Investigation (Lab) AEs | 6 | 3 | 23
  Metabolism and Nutrition AEs | 5 | 2 | 45
  Musculoskeletal and Connective Tissue AEs | 4 | 1 | 2
  Nervous System AEs | 13 | 3 | 5
  Renal and Urinary AEs | 0 | 1 | 4
  Reproductive System AEs | 0 | 1 | 1
  Respiratory, thoracic and mediastinal AEs | 10 | 4 | 15
  Skin and Subcutaneous Tissue AEs | 8 | 2 | 3
  Vascular AEs | 2 | 1 | 1

4. Secondary Outcome: Distribution of Change Across Time of mTOR and HDAC-I Inhibition From Baseline Until After the 1st 2 Cycles of Study Drug in Patients Who Received LBH and RAD.
Description: Serum markers will be measured on the first day of cycle 1 and on the first day of cycle 3. The distribution of change across time in a marker will be summarized.
Time Frame: after 2 cycles of study therapy; up to 8 weeks
Population: The number of responses to treatment were so few that we did not think we could get enough meaningful data for analysis. Therefore, serum marker analysis was not performed and no results are available.
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Evaluate the Association of Observed Response to the Doublet With the Response Predicted by Molecular Signatures for Activated B Cell Like (ABC) DLBCL and for Germinal Center B Cell Like (GCB) DLBCL.
Description: Response rates seen in subjects with activated B cell like DLBCL and for Germinal center B cell like DLBCL will be reported and assessed to see if GCB is associated with improved outcomes compared to ABC in subjects with relapsed disease who have received RAD + LBH. We will estimate the association of the ABC and GCB with the observed response. All evaluable patients will be used in estimating response. The chi-square test with one-sided alpha of 0.10 will be used to test for the association between predicted and observed responses.
  The number of responses to treatment were so few that we did not think we could get enough meaningful data for analysis.
Time Frame: up to 13 cycles of therapy; approximately 1 year
Population: as for outcome 2
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of consent until 4 weeks after the last dose of study drug; approximately 1 year.
Arm/Group | Arm 1a (RAD001 Followed by LBH589) | Arm 1b (LBH589 Followed by RAD001) | Doublet (Combination RAD001 and LBH589)
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/5 | 6/18
Other Adverse Events (participants affected / at risk) | 10/10 | 5/5 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1a (RAD001 Followed by LBH589) (N=10) | Arm 1b (LBH589 Followed by RAD001) (N=5) | Doublet (Combination RAD001 and LBH589) (N=18)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 1a (RAD001 Followed by LBH589) (N=10) | Arm 1b (LBH589 Followed by RAD001) (N=5) | Doublet (Combination RAD001 and LBH589) (N=18)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 9 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 4 (4) | 15 (21)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 5 (8) | 2 (2) | 12 (16)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal - Other (Burping) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other (Gas) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (1) | 4 (5)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4/5 (5) | 1 (1) | 3 (3)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 3 (4)
Fatigue (General disorders) | 4 (4) | 3 (3) | 12 (14)
Non-cardiac Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Infections and Infestations - Other (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Cholesterol high (Investigations) | 2 (2) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 2 (3) | 2 (2) | 5 (7)
Weight loss (Investigations) | 1 (1) | 1 (1) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (5) | 1 (1) | 3 (3)
Dysphagia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other (Dry Throat) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Rash, NOS) (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes